CLINICAL TRIAL: NCT01124565
Title: A Phase 2, Open-Label, Repeat Dose, Multi-Center Study to Evaluate the Safety of RT001 Topical Gel for the Treatment of Moderate to Severe Lateral Canthal Lines in Adults
Brief Title: Safety Study of Two Repeat Doses of RT001 for the Treatment of Moderate to Severe Lateral Canthal Lines in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT001-CL025LCL
Record Dates: First submitted 2010-05-12; First posted 2010-05-17 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2013-12

CONDITIONS: Lateral Canthal Lines; Crow's Feet; Facial Wrinkles
Keywords: Lateral Canthal Lines; Crow's Feet; Facial Wrinkles
MeSH Terms: interventions — RT001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RT001 (Experimental): RT001 (Botulinum Toxin Type A) Topical Gel
  Interventions: Drug: RT001

INTERVENTIONS:
Drug: RT001 — RT001 (Botulinum Toxin Type A Topical Gel, Dose A) at Baseline (Day 0) and Week 4 to the lateral canthal areas

SUMMARY:
This study's objective is to evaluate if RT001 is safe and well-tolerated following two (2) sequential applications.

DETAILED DESCRIPTION:
Revance is conducting this Phase 2 clinical study to establish the safety of two (2) sequential doses of RT001 Topical Gel at Baseline (Day 0) and Week 4 for the treatment of moderate to severe LCLs at rest.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent including authorization to release health information
* Female or male, 18 to 65 years of age and in good general health
* Willing and able to follow study instructions and likely to complete all study requirements
* Moderate to severe lateral canthal lines (crow's feet wrinkles)

Exclusion Criteria:

* Any neurological condition that may place the subject at increased risk with exposure to Botulinum Toxin Type A, including peripheral motor neuropathic diseases such as amyotrophic lateral sclerosis and motor neuropathy, and neuromuscular junctional disorders such as Lambert-Eaton syndrome and myasthenia gravis
* Muscle weakness or paralysis, particularly in the area receiving study treatment
* Active disease or irritation at the treatment areas including the eye and the skin
* Pregnant, nursing, or planning a pregnancy during the study; or is a woman of child bearing potential (WOCBP) but is not willing to use an effective method of birth control
* Previous participation in a RT001 clinical study
* Previous treatment with botulinum toxin (any serotype)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Assessment of treatment-emergent adverse events based on safety assessments. | 4 weeks and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joel Schlessinger, M.D., Principal Investigator — Skin Specialists, PC
Locations (3):
- United States (3):
  - Total Skin & Beauty Dermatology Center, PC, Birmingham, Alabama
  - Therapeutics Clinical Research, San Diego, California
  - Skin Specialists, PC, Omaha, Nebraska